CLINICAL TRIAL: NCT05774912
Title: Fetal Growth Curves and Doppler Velocimetry in the Italian Population, Multicenter Study
Brief Title: Development of Italian Fetal Growth Charts
Acronym: METRICS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 24/20
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2023-06

CONDITIONS: Growth Charts
Keywords: Fetal growth charts; Doppler; biometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Healthy women with singleton uncomplicated pregnancy
  Interventions: Other: Ultrasound evaluation

INTERVENTIONS:
Other: Ultrasound evaluation — Fetal ultrasound evaluation will be collected longitudinally during the prenatal period from the weeks 14 every 4-5 weeks, for a total of maximum 6 ultrasound scans

SUMMARY:
There is an ongoing international discussion regarding which fetal growth charts should be used. As a matter of fact, an extensive and clinically significant variability among different growth charts has been proved, even between studies of the highest methodological quality. Indeed, methodological aspects such as the study population, data collection, curve modeling and others are of crucial importance for the final outcome of the process. Beside the discussion on methodological issues, there is also an ongoing discussion regarding whether one international standard might be adequate to assess fetal growth all around the globe, or are there some differences related to ethnicity supporting the adoption of growth charts constructed based on national data, or even the customization. Recently, the International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) Practice Guidelines on Ultrasound Assessment of Fetal Biometry and Growth recommended the application of "prescriptive biometry charts, obtained prospectively, truly population-based and derived from studies with the lowest possible methodological bias", and called for the practitioners' awareness regarding national or even local reference charts. Such awareness requires an exploratory and preliminary analysis of the impact of different charts by applying reference values to local findings.

On these grounds, there is an urgent need for a nationwide study for the prospective collection of data and the construction of methodologically robust national growth and Doppler standards.

DETAILED DESCRIPTION:
There is an ongoing international discussion regarding which fetal growth charts should be used. As a matter of fact, an extensive and clinically significant variability among different growth charts has been proved, even between studies of the highest methodological quality. Indeed, methodological aspects such as the study population, data collection, curve modeling and others are of crucial importance for the final outcome of the process. Beside the discussion on methodological issues, there is also an ongoing discussion regarding whether one international standard might be adequate to assess fetal growth all around the globe, or are there some differences related to ethnicity supporting the adoption of growth charts constructed based on national data, or even the customization.

Recently, the International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) Practice Guidelines on Ultrasound Assessment of Fetal Biometry and Growth recommended the application of "prescriptive biometry charts, obtained prospectively, truly population-based and derived from studies with the lowest possible methodological bias", and called for the practitioners' awareness regarding national or even local reference charts. Such awareness requires an exploratory and preliminary analysis of the impact of different charts by applying reference values to local findings.

A recent multicentric Italian study promoted by the Italian Society of Ultrasound in Obstetrics and Gynecology (SIEOG), assessed the application of WHO growth charts published in 2006 and the Intergrowth 21 (IG-21st) growth charts in a large Italian cohort (n=7347) of low risk women with uneventful pregnancy. According to the results of the study the IG-21st standards identified the smallest proportion of fetuses below the 10th centile and the largest proportion of fetuses above the 90th centile, respectively. The proportion of fetuses with head circumference (HC), abdominal circumference (AC) and femur length (LF) above 90th centile was 29.9%, 32.5 and 46%, respectively. While the WHO references seem to be the closest to observed 10th centile, the proportion of fetuses above 90th centile was also higher than expected for an appropriate distribution of centiles, but smaller compared with IG-21st standards: 22.8%, 21.3% and 31.9% for HC, AC and LF, respectively. Overall, these data suggest that there might be differences linked to ethnic origin and not fully explained by maternal, socio-economic or other methodological factors as already suggested by the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) and World Health Organization (WHO) groups.

These data suggest that, despite indisputable advantages that IG-21st growth standards might offer, immediate application into clinical practice might result into an under-diagnosis of small for gestational age fetuses and, especially, in an over-diagnosis of large for gestational age fetuses with major consequences for clinical practice. The WHO growth references seem to be more suitable for our population, although they might also over-estimate the proportion of large for gestational age fetuses. On the other hand, existing national growth charts lack crucial biometric parameters and centiles. This is of major importance, if we consider that recent consensus criteria suggested AC and estimated fetal weight (EFW) below the 3rd centile as independent criteria for the diagnosis fetal growth restriction.

On these grounds, there is an urgent need for a nationwide study for the prospective collection of data and the construction of methodologically robust national growth and Doppler standards.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years and ≤40 years
2. body mass index (BMI) 18-30 kg/m2
3. singleton pregnancy
4. the first day of the last menstrual period (LMP) known and the cycle reported to be regular, lasting 28 days ±4 days and a crown rump length (CRL) measured in early pregnancy
5. no history of chronic health problems
6. no long-term medication (including fertility treatment)
7. no environmental or economic constraints likely to impede fetal growth
8. not smoking currently or in the previous 6 months
9. no alcohol consumption
10. no history of recurrent miscarriages
11. no previous preterm delivery (<37 week) or birthweight < 2,500 grams
12. no evidence in the present pregnancy of congenital disease or fetal anomaly at study entry

Exclusion Criteria:

1. multiple pregnancy
2. fetuses with congenital structural or chromosomal anomalies including increased nuchal translucency (>99°centile)
3. fetal death
4. women with disorders that may affect fetal growth (pre-existing hypertension, diabetes mellitus, renal disease)
5. drug assumption (low dose aspirin, etc)
6. smoking
7. delivery <37 weeks
8. pregnancy complications (hypertensive disorders of pregnancy, infections, gestational diabetes, other diseases)
9. pregnancies conceived by assisted reproductive technology
10. Abnormal uterine arteries Doppler (if performed)
11. First trimester PAPP-A<0.3 MoM

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Healthy women with singleton uncomplicated pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Fetal growth evaluation | From the weeks 14 of gestational age to delivery
  Construction of national normal fetal growth reference charts

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Stampalija, Study Chair — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (3):
- Italy (3):
  - Fondazione Policlinico Agostino Gemelli - IRCCS City Rome, Rome, Lazio
  - Fondazione IRCSS Ca Granda, Policlinico di Milano, Milan, Lombardy
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste

IPD SHARING:
Plan to Share IPD: Undecided